CLINICAL TRIAL: NCT02711280
Title: The Effect of Sevoflurane and Propofol on Oxidative Stress and Apoptosis Status in Children Undergoing Hypospadias Repair Surgery
Brief Title: The Effect of Anesthetics on Oxidative Stress and Apoptosis Status in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Feng Xia, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: [2014]114
Record Dates: First submitted 2016-03-07; First posted 2016-03-17 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Sevoflurane General anesthesia (Experimental): Anesthesia was induced with 8% sevoflurane with 8L/min oxygen. Anesthesia was maintained with 1-3% sevoflurane in oxygen/air mixture.
  Interventions: Drug: Sevoflurane
- Propofol General anesthesia (Experimental): Anesthesia was induced with propofol 4mg/kg. Anesthesia was maintained with propofol 7-12mg/kg/h.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane
  Arms: Sevoflurane General anesthesia
Drug: Propofol
  Arms: Propofol General anesthesia

SUMMARY:
The purpose of this study is to determine whether Propofol and Sevoflurane affect the oxidative stress and apoptosis status in children undergoing hypospadias repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I-II, undergoing selective surgery for hypospadias repair.

Exclusion Criteria:

* a history of developmental delay or mental retardation, which could make observational pain intensity assessment outside the norm;
* a history of central nervous system diseases;
* a known or suspected coagulopathy;
* a known allergy to any of the study drugs;
* abnormalities of the sacrum and any signs of infection at the site of the proposed caudal block.

Ages: 1 Year to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
the change of blood glutathione peroxidase(GPx) level in perioperative period | immediately after anesthetic induction, 2h and 3 days after operation
the change of blood-separated erythrocytes superoxide dismutase (SOD) activities in perioperative period | immediately after anesthetic induction, 2h and 3 days after operation
  the blood sample was separated and erythrocytes was obtained, superoxide dismutase activity was measured using a commercially available assay-Ransod kit (Randox Laboratories, UK).
the change of blood-separated erythrocytes catalase (CAT) activities in perioperative period | immediately after anesthetic induction, 2h and 3 days after operation
  the blood sample was separated and erythrocytes was obtained, catalase activity was measured using the OxiSelect catalase activity assay (Cell Biolabs, San Diego, CA, USA)
the change of blood-separated lymphocytes caspase-3 mRNA level in perioperative period | immediately after anesthetic induction, 2h and 3 days after operation
  Lymphocytes were separated from whole blood and freshly used for real-time PCR of caspase-3

CONTACTS AND LOCATIONS:
Overall Officials: Xue Zhou, Master, Principal Investigator — Department of Anesthesiology, the First-Affiliated Hospital of Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China